CLINICAL TRIAL: NCT05509218
Title: Daily Personalized Drinking Feedback Delivered Via Mobile Phone
Brief Title: Alcohol Feedback, Reflection and Morning Evaluation
Acronym: (A-FRAME)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022003299; 1R34AA029733-01A1 (NIH)
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Youth Drinking; Alcohol Drinking
Keywords: young adults; personalized feedback intervention; mobile intervention; alcohol use
MeSH Terms: conditions — Underage Drinking; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of three conditions: (1) daily surveys plus personalized feedback about yesterday's drinking, with a monetary incentive for survey completion, (2) daily surveys plus personalized feedback about yesterday's drinking, with no monetary incentive, or (3) survey assessment (baseline and follow-up) only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized feedback plus incentive (Experimental): Following each daily survey on which a participant indicates prior day drinking, personalized feedback will be provided. Participants in this group will receive $1 per day for submitting their daily survey.
  Interventions: Behavioral: Mobile-delivered personalized feedback
- Personalized feedback without incentive (Experimental): Following each daily survey on which a participant indicates prior day drinking, personalized feedback will be provided. Participants in this group will NOT receive $1 per day for submitting their daily survey.
  Interventions: Behavioral: Mobile-delivered personalized feedback
- Control (No Intervention): Participants in this arm will only complete baseline and follow-up surveys.

INTERVENTIONS:
Behavioral: Mobile-delivered personalized feedback — Following each daily survey on which a participant indicates prior day drinking, personalized feedback will be provided on how their most recent behavior (e.g., drinks last night, drinking days so far this week) compare/contrast with personal goals. Participants will then choose whether to receive additional feedback in any of 7 areas: blood alcohol concentrate on, high risk behaviors, consequences of drinking, caloric intake, spending, how drinking compares to peers, and safe drinking strategies. All participants will receive feedback on drinks consumed, and then be asked to choose at least one additional topic for feedback (following each drinking day). In addition to day-level feedback, an aggregate feedback report on drinking patterns and related behaviors will be delivered twice, once at the end of each 2-week period. Once again, they will have the option to view feedback across the range of topics noted above.
  Arms: Personalized feedback plus incentive; Personalized feedback without incentive

SUMMARY:
The investigators propose to examine mornings after drinking as an optimal time to provide repeated, personalized feedback, with the goal of reducing hazardous drinking. Specifically, the investigators will further develop and pilot test a novel theory-based personalized feedback intervention (PFI) for heavy drinking young adults. Intervention strategies include personalized feedback (e.g., feedback on prior night blood alcohol concentration, consequences) contrasted with both drinking goals set at baseline and corrective normative feedback (e.g., how last night's drinking compares to peers). Up to 170 participants (50% non-college) will be randomized to one of three groups: PFI with monetary incentives for daily surveys, PFI without monetary incentives, or survey assessment only. The investigators will examine recruitment rates, retention rates, confirmation of intervention content delivery/intake, response rates to daily surveys, data quality, and ratings of intervention value. Investigators will test whether these indicators of engagement differ between those who do and do not receive monetary incentives for daily surveys. Further, baseline, post-test, and 3-month follow-up assessments will allow us to examine differences in drinking behavior between PFI and control. The results of the proposed research will result in a novel and scalable intervention for alcohol misuse among young adults, with potential to have an important impact on the public health problem of high-risk drinking.

DETAILED DESCRIPTION:
The investigators will recruit up to 170 participants for a small randomized controlled trial. Participants will be randomized to four weeks of intervention with or without daily incentives for completing surveys, or assessment-only control, to test feasibility, acceptability, and initial evidence of efficacy.

1. Baseline assessment and orientation. An orientation meeting will be used to describe all study procedures and obtain informed consent. If informed consent is obtained, participants will then be given one week to complete a baseline survey (~30 minutes) on their own time, using their own computers. Data needed to personalize the intervention content will be collected during the baseline survey. Participants will be asked to choose from a range of possible goal types (e.g., max drinks per drinking event, drinks per week, weekly frequency of drinking, "skip goals", "delay goals", slow goals", "stop goals"). These goals an be integrated/contrasted with subsequent self-reported behavior on morning reports during the intervention period. After the baseline survey, a research assistant (RA) will review study procedures.
2. Randomization. Randomization will occur following consent. The pilot randomized controlled trial (RCT) will include three conditions (mobile PFI with daily incentive for surveys, mobile PFI without daily incentives, assessment-only). PFI participants (both groups) will also complete (1) orientation and participant training (as described above), (2) four weeks of daily assessment and (3) intervention (as described below), and (4) follow-up surveys.
3. Daily assessment. Daily assessment + feedback will begin on a Monday for all participants. A link to a web-based morning survey will be sent at 7am, and it will remain available until 2pm. When prior night alcohol use is endorsed, details will be assessed via single item measures about the drinking event.
4. Personalized Feedback Reports. Following each daily survey on which a participant (in PFI groups) indicates prior day drinking, personalized feedback will be provided on how their most recent behavior (e.g., drinks last night, drinking days so far this week) compare/contrast with personal goals. Participants will then choose whether to receive additional feedback in any of 7 areas: blood alcohol concentration, high risk behaviors, consequences of drinking, caloric intake, spending, how drinking compares to peers, and safe drinking strategies. In addition to day-level feedback, an aggregate feedback report on drinking patterns and related behaviors will be delivered twice, once at the end of each 2-week period. At the end of the 2-week feedback report, participants in the intervention groups will have the opportunity to update/add goals for the next 2 weeks, given what they learned thus far about their personalized behavior-outcome links.
5. Follow-up surveys. At the end of four weeks, participants in all three groups will complete a 30-minute online survey (post-intervention). The final 30-minute follow-up will take place three months after the end of intervention (four months after baseline) and will assess primary outcomes and mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-29 years
* Own a smartphone and use it daily
* Heavy episodic drinking (4+/5+ drinks for women/men) at least weekly in past month
* At least one of 10 negative consequences assessed
* at least somewhat willing to consider drinking even a little less than current

Exclusion Criteria:

* current participation in treatment for an alcohol or other substance use disorder
* participation in an earlier phase of the study
* enrollment in ongoing alcohol studies at the same university

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
drinks per week | post-test (end of 4-week intervention) and 3-month follow-up (3 months after end of intervention)
  Number of drinks consumed per typical week in the past 30 days
heavy drinking frequency | post-test (end of 4-week intervention) and 3-month follow-up (3 months after end of intervention)
  Number of days drinking 4+ drinks (women) or 5+ drinks (men) in the past 30 days
negative alcohol consequences | post-test (end of 4-week intervention) and 3-month follow-up (3 months after end of intervention)
  Number of consequences reported on the 24-item Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Merrill, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit and share data with NIAAA Data Archive, a data repository housed within the National Institute of Mental Health Data Archive (NDA). Participants complete a baseline survey of participant characteristics and drinking behavior and related constructs, a post-test survey, and a 3-month follow-up assessment to measure drinking behavior post-intervention. Data from these 3 surveys will be shared.
Time Frame: Data will be shared on or before the NDA submission due dates (April 1 and October 1 each year). It will remain in the archive as per the archive regulations.